CLINICAL TRIAL: NCT01994590
Title: A Phase II Study of Dovitinib (TKI258) Combined With Abiraterone Acetate in Patients With Metastatic Castrate-Resistant Prostate Cancer Evaluating Markers of FGF and AR Signaling in Bone Marrow and Plasma
Brief Title: Dovitinib (TKI258) and Abiraterone Acetate in Metastatic Castrate-Resistant Prostate Cancer (mCRPC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor stopped supplying study drug
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0086; NCI-2014-00887 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-11-19; First posted 2013-11-26 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Metastatic Castrate-Resistant Prostate Cancer; mCRPC; Dovitinib; TKI258; Abiraterone Acetate; Zytiga; Prednisone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dovitinib + Abiraterone Acetate + Prednisone (Experimental): Participants receive a single daily oral dose of Dovitinib for 5 consecutive days, on Days 1-5, 8-12, 15-19, and 22-26 of each 28 day cycle. Starting dose will be 400 mg daily.
  Participant to take 4 tablets (250 mg each) orally (PO) daily of Abiraterone acetate.
  Participant to take 5 mg oral prednisone, twice daily.
  Interventions: Drug: Dovitinib; Drug: Abiraterone Acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Dovitinib — Starting dose will be 400 mg by mouth daily on Days 1-5, 8-12, 15-19, and 22-26 of each 28 day cycle.
  Other Names: TKI258
Drug: Abiraterone Acetate — 4 tablets (250 mg each) by mouth daily.
  Other Names: Zytiga
Drug: Prednisone — 5 mg by mouth twice daily.

SUMMARY:
The goal of this clinical research study is to learn if adding dovitinib to the combination of abiraterone acetate and prednisone may help to control metastatic CRPC. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will take the study drugs in 28-day cycles.

Dovitinib:

You will take dovitinib capsules by mouth 1 time each day on Days 1-5, 8-12, 15-19, and 22-26 of each cycle. You should take the dovitinib with about a cup (8 ounces) of water. You may take dovitinib with or without food.

If you miss a dose of dovitinib on Days 1-4, 8-11, 15-18, or 22-25, you should not make up the dose on the same day. You should continue taking the drug as scheduled the following day.

If you miss a dose on Days 5, 12, 19, or 26, you should skip the dose, wait 2 days, and start taking dovitinib again as scheduled (on Day 8, 15, 22, or 1 of the next cycle). The study doctor will talk to you about what else you need to do if you miss a dose.

Abiraterone Acetate:

You will take 4 abiraterone acetate tablets by mouth 1 time each day at least 1 hour before a meal or 2 hours after a meal. You should take the abiraterone acetate tablets at about the same time each day and swallow them whole with water. Do not crush or chew the abiraterone acetate tablets.

Prednisone:

You will take 1 tablet of prednisone by mouth 2 times each day (once in the morning, and once in the evening) to help lower the risk of side effects caused by abiraterone acetate.

You should return all unused study drug and/or empty pill bottles to the clinic at the end of each cycle.

If you have side effects, the study doctor may lower the dose of dovitinib and/or abiraterone acetate.

Study Visits:

On Day 1 of every cycle:

* You will have a physical exam.
* Blood (about 3 tablespoons) will be drawn for routine tests, to check your prostatic specific antigen (PSA) levels, and to check how well your blood clots. You must fast for at least 8 hours before this blood draw. On Day 1 of Cycles 2 and 3 only, this blood will also be used for biomarker testing.
* Urine will be collected for routine tests.

On Day 1 of Cycles 1 and 2, and then every odd-numbered cycle afterward (Cycles 3, 5, 7, and so on):

* Blood (about 2 teaspoons) will be drawn for routine tests.
* Urine will be collected to test for markers relating to your bone.

On Day 1 of Cycles 1-3, you will have an EKG.

On Day 1 of Cycle 1, and then on Day 1 of every 3 cycles (Cycles 4, 7, 10, and so on), blood (about 1 tablespoon) will be drawn to test your thyroid function.

On Day 14 of Cycle 1:

* You will have a physical exam.
* Blood (about 3 tablespoons) will be drawn for routine tests and to check how well your blood clots. You must fast for at least 8 hours before this blood draw.
* Urine will be collected for routine tests.

On Day 14 of Cycles 2 and 3, blood (about 1 tablespoon) will be drawn for routine tests.

Every 8 weeks for the first 6 months and every 3 months after that, you will have a chest x-ray, bone scan, and either a CT or MRI scan of your abdomen and pelvis to check the status of the disease.

About 7-10 weeks after your first dose of study drug, you will have another bone marrow biopsy and aspiration performed to check the status of the disease and for biomarker testing.

At Weeks 12 and 24, you will have an echocardiogram or MUGA scan.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You may no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

End-of-Treatment Visit:

Within 4 weeks after your last dose of the study drugs, you will return to the clinic for an end-of-treatment visit. The following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 3 tablespoons) will be drawn for routine tests and to check your PSA levels. This blood will also be used for biomarker testing. You will need to fast for at least 8 hours before this blood draw.
* Urine will be collected to test for markers relating to your bone. You will have a chest x-ray, bone scan, CT scan, and/or MRI of your abdomen and pelvis to check the status of the disease.
* You will have an EKG and either an echocardiogram or a MUGA scan to check your heart function.
* You will have a bone marrow biopsy and aspiration performed to check the status of the disease and for biomarker testing.

Long-Term Follow-up:

The study staff will check up on you to ask how you are doing about every 3 months after your end-of-treatment visit. This update will consist of a phone call, an e-mail, or clinic visit. If contacted by phone, the call would last about 5 minutes.

This is an investigational study. Dovitinib is not FDA approved or commercially available. It is currently being used for research purposes only.

Abiraterone acetate is FDA approved in combination with prednisone for the treatment of metastatic CRPC in patients who have received docetaxel. Its use in this study is investigational.

Prednisone is FDA approved and commercially available as a corticosteroid. It is commonly used with abiraterone acetate.

The study doctor can explain how the study drugs are designed to work.

Up to 60 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or his legally authorized representative must provide written informed consent.
2. Age >/= 18
3. Eastern Cooperative Oncology Group (ECOG) performance status </= 2
4. Histologic evidence of prostate adenocarcinoma
5. Diagnosis of metastatic castration-resistant prostate cancer, with measureable disease (lymph nodes and/or visceral metastases by RECIST) or bone metastases.
6. Patients must have surgical or ongoing chemical castration (with LHRH agonists or LHRH antagonists), with a baseline testosterone level < 50ng/dL
7. Patients must have documented evidence of progressive disease as defined by any of the following: a) PSA progression: minimum of 2 rising values (3 measurements) obtained a minimum of 7 days apart with the last result being at least >/= 2.0 ng/mL; b) New or increasing non-bone disease (RECIST); c) A positive bone scan with 2 or more new lesions (PCWG2). Patients must have evidence for metastatic prostate cancer by bone scan and/or CT/MRI (i.e., soft tissue, visceral, lymph node). If lymph node, visceral and/or soft-tissue metastases are the only evidence of metastasis, at least one lesion must be >/= 1.5 cm in diameter.
8. Laboratory requirements: a) Absolute neutrophil count (ANC) >/= 1,500/ml; b) Platelets >/= 100,000/ml; c) Total bilirubin </= 1.5 x upper limit of normal (ULN); d) Serum glutamate pyruvate transaminase (SGPT) (ALT) AND/OR Serum glutamate oxaloacetate transaminase (SGOT) (AST) </= 3.0 x ULN; e) Creatinine </= 1.5 x ULN; f) White blood cell count (WBC) >/= 3,000 uL; g) Hb >/= 8.0 g/dL independent of transfusion
9. Men whose partner is a woman of childbearing potential must be willing to consent to using effective contraception (e.g. male condom with spermicide, diaphragm with spermicide, intra-uterine device) while on treatment and for at least 3 months thereafter.
10. Patients may have received prior treatment with androgen ablative therapies (e.g. bicalutamide, DES, enzalutamide) and/or "targeted" therapies (such as tyrosine kinase inhibitors). Androgen ablative therapies must be discontinued >/=3 days prior to initiation of study treatment with the exception of enzalutamide which may be continued during protocol treatment per the practice preference of the treating physician. Patients who are predicted to benefit from an antiandrogen withdrawal response should be tested for this possibility before being considered for eligibility to this study. Targeted therapies must be discontinued >/= 2 weeks before initiation of study treatment.
11. Patients may have received up to 2 prior cytotoxic chemotherapy regimens for the treatment of metastatic castration-resistant disease, but these therapies must be discontinued >/= 3weeks before initiation of study treatment. At least one of the regimens must have contained docetaxel and patients must have recovered to < Grade 2 adverse events from prior chemotherapy or to pretreatment baseline

Exclusion Criteria:

1. Patients with histologic evidence of small cell carcinoma of the prostate
2. Prior therapy with dovitinib or abiraterone acetate or other FGF targeted therapy
3. Radiation therapy (including palliative radiotherapy to a metastatic lesion) within 14 days
4. Major surgery (e.g., open abdominal, pelvic, thoracic, orthopedic or neurosurgery) within 28 days of the date of the first dose of study drugs
5. Samarium-153 within 28 days of the date of the first dose of study drugs, or Strontium-89 within 12 weeks (84 days) of the date of the first dose of study drugs. Patients who have received 2 or more doses of bone-seeking radioisotopes are not eligible
6. Current treatment on another therapeutic clinical trial
7. Impending complication from bone metastases (fracture and/or cord compression). Properly treated or stabilized fractures and/or cord compression is allowed
8. Presence of ongoing urinary obstruction (e.g., urinary retention, hydronephrosis) requiring medical intervention. Urinary obstruction relieved with treatment is allowed
9. Patient has an uncontrolled intercurrent illness (e.g., uncontrolled diabetes, uncontrolled hypertension)
10. Patient has another serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the patient's ability to provide informed consent or with the completion of treatment according to this protocol
11. Patients with an active second malignancy that could, in the investigator's opinion, potentially interfere with the patient's ability to participate and/or complete this trial
12. Patients with known brain metastases
13. Impaired cardiac function or clinically significant cardiac diseases, including any of the following: a.) History or presence of serious uncontrolled ventricular arrhythmias; b. Clinically significant resting bradycardia; c.) Left ventricular ejection fraction (LVEF) assessed by 2-D echocardiogram (ECHO) < 50% or lower limit of normal (whichever is the higher), or 2-D multiple gated acquisition scan (MUGA) < 45% or lower limit of normal (whichever is the higher); d.) Any of the following within 6 months prior to starting study drug: myocardial infarction (MI), severe/unstable angina, Coronary Artery Bypass Graft (CABG), Congestive Heart Failure (CHF), Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA);
14. (Exclusion #14 continued) e.) Chronically uncontrolled hypertension, defined conventionally as consistent/repeated systolic pressures above 140 mmHg or diastolic pressures above 90 mmHg despite anti-hypertensive therapy. This may be established with home BP readings. There is no criterion related to a specific BP result required for eligibility, nor are acute BP elevations that are related to iatrogenic causes, acute pain, or other transient reversible causes considered an exclusion criterion. The intent is to exclude patients with chronically uncontrolled hypertension that might be further exacerbated by the study drugs.
15. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of dovitinib (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or gastric or small bowel resection)
16. Cirrhosis, chronic active hepatitis or chronic persistent hepatitis
17. Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory) or hepatitis B virus (HBV) or hepatitis C virus (HCV) disease or antigen positivity
18. Initiation of bisphosphonate and/or RANKL inhibitors within 4 weeks prior to first dose of study drug. Patients already on stable doses of bisphosphonates and/or RANKL inhibitors may continue these drugs. However, patients are not allowed to initiate bisphosphonate and/or RANKL inhibitors during the study
19. Any bleeding dyscrasia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-05-19 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Corn, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Dovitinib combined with abiraterone and prednisone
Period: Overall Study
Arm/Group | All Patients
Started | 4
Completed | 2
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Trial Terminated | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 71.25 [66 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Number of Participants with Adverse Events
Time Frame: Participants are followed while actively taking study drug and for at least 30 days post last dose.
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: First study drug dose, until 30 days after the last dose of study drug, unless the participant withdraws consent
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=4)
Thromboembolic Event (Blood and lymphatic system disorders) | 1
Skin Infection (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=4)
Alanine aminotransferase increased (Hepatobiliary disorders) | 2
Alkaline phophatase increased (Hepatobiliary disorders) | 2
Anemia (Blood and lymphatic system disorders) | 2
Aspartate aminotransferase increase (Hepatobiliary disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (Metabolism and nutrition disorders) | 4
Hematuria (Renal and urinary disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesium (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 1
Localized edema (Blood and lymphatic system disorders) | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 3
Proteinuria (Renal and urinary disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2
Urinary tract infection (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
White blood cell decreased (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT01994590/Prot_SAP_000.pdf